CLINICAL TRIAL: NCT00454558
Title: A Multicenter, Non-randomized, Non-blinded, Noncontrolled Study to Investigate the Impact of Multiple Doses of BAY 63-2521 on Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics in Patients With Pulmonary Hypertension in a 12-week 3 Times a Day Individual Dose Titration Scheme
Brief Title: An Open Multiple Dose Titration Study In Patients With Pulmonary Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12166; 2006-003520-10 (EudraCT Number)
Record Dates: First submitted 2007-03-28; First posted 2007-03-30 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-09

CONDITIONS: Hypertension, Pulmonary
Keywords: Pulmonary Arterial Hypertension (PAH); Chronic Thromboembolic Pulmonary Hypertension (CTEPH)
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — riociguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Riociguat (Adempas, BAY63-2521)

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY63-2521) — Biweekly uptitration of BAY63-2521 (Oral sGC Stimulator) starting from 1.0 mg TID up to 2.5 mg TID in steps of +0.5 mg according to safety and tolerability.

SUMMARY:
This is a study to demonstrate the feasibility of an individual dose titration scheme based on the systolic blood pressure with a dose range from 1.0 mg TID to 2.5 mg TID. Patients suffering from chronic thromboembolic pulmonary hypertension (CTEPH) or pulmonary arterial hypertension (PAH) will be included. After diagnosis by an expert center, patients receive medication three times a day starting with 1.0 mg TID. The first tablets are given in the hospital, then the patients are allowed to go home and take the medication at home. After 2 weeks, patients return to the hospital for an ambulatory visit and the dose may be increased based on the actual condition of the patient (blood pressure and adverse events). Several measurements will be performed to test the efficacy of the drug and whether there are any unwanted reactions to the drug (blood tests, ECG, 6 minute walk test, imaging by Echo, quality of life scores). The dose of the drug will then be increased further until unwanted effects may occur or the blood pressure drops to low. The highest dose tested will be 2.5 mg TID. After 12 weeks the patient is going to stay in the hospital again and a right heart catheter is performed to examine the changes in hemodynamics after 12 weeks of treatment with the drug. If the patients give their consent they can enter a long-term extension trial continuing on BAY63-2521 with the dose reached after 12 weeks. Every 3 months an ambulatory visit at the specialist center will be performed including measurements of safety (blood tests, ECG, clinical assessment) and efficacy (6 minute walk test, Borg dyspnea scale, NT-pro BNP). Blood tests and ECG have been removed begin of 2013 as safety parameter by amendment 7; furthermore Borg dyspnea score and NT-proBNP have been removed as efficacy parameter.

Initially the inclusion of ten patients suffering from chronic thromboembolic pulmonary hypertension (CTEPH) or pulmonary arterial hypertension (PAH) was planned. Later on the patient number was amended and 75 patients entered the trial.

Furthermore the trial duration was extended and a long term treatment with BAY63-2521 was offered to the patients. Finally 68 patients moved over to the long term extension period of the trial.

DETAILED DESCRIPTION:
Specification of primary outcome measures for long-term safety and tolerability: Adverse events, blood pressure and heart rate, 12 lead ECG, clinical chemistry and hematology, Troponin I

ELIGIBILITY:
Inclusion Criteria:

* Patients with CTEPH or PAH in NYHA class II or III

Exclusion Criteria:

* Patients with PDE 5 inhibitor or prostacycline pretreatment, relevant pulmonary diseases, relevant cardiac diseases, severe coagulation disorders, moderate to severe hepatic or renal insufficiency, pregnancy, hypotension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-01; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
To investigate the safety, tolerability and feasibility of individual titration of BAY63-2521 according to peripheral systolic blood pressure | 3 months
To investigate the long term safety and tolerability of BAY63-2521 | max. 84 months

SECONDARY OUTCOMES:
6MWT | max. 84 months
Right heart catheter invasive hemodynamics | 3 months
WHO functional class assessment | max. 84 months
NT-pro BNP | 75 months
Imaging by echo | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (15):
- Germany (15):
  - Heidelberg, Baden-Wurttemberg
  - Löwenstein, Baden-Wurttemberg
  - München, Bavaria
  - Regensburg, Bavaria
  - Hamburg, Hamburg
  - Bad Nauheim, Hesse
  - Giessen, Hesse
  - Hanover, Lower Saxony
  - Greifswald, Mecklenburg-Vorpommern
  - Cologne, North Rhine-Westphalia
  - Homburg, Saarland
  - Dresden, Saxony
  - Leipzig, Saxony
  - Halle, Saxony-Anhalt
  - Berlin, State of Berlin

REFERENCES:
- [Result] Belik J. Riociguat, an oral soluble guanylate cyclase stimulator for the treatment of pulmonary hypertension. Curr Opin Investig Drugs. 2009 Sep;10(9):971-9. PMID 19705340
- [Result] Ghofrani HA, Hoeper MM, Halank M, Meyer FJ, Staehler G, Behr J, Ewert R, Weimann G, Grimminger F. Riociguat for chronic thromboembolic pulmonary hypertension and pulmonary arterial hypertension: a phase II study. Eur Respir J. 2010 Oct;36(4):792-9. doi: 10.1183/09031936.00182909. Epub 2010 Jun 7. PMID 20530034
- [Derived] Halank M, Hoeper MM, Ghofrani HA, Meyer FJ, Stahler G, Behr J, Ewert R, Fletcher M, Colorado P, Nikkho S, Grimminger F. Riociguat for pulmonary arterial hypertension and chronic thromboembolic pulmonary hypertension: Results from a phase II long-term extension study. Respir Med. 2017 Jul;128:50-56. doi: 10.1016/j.rmed.2017.05.008. Epub 2017 May 16. PMID 28610669